CLINICAL TRIAL: NCT00282165
Title: Efficacy of a Triptan in the Treatment of Hostility and Aggression Among Convicts With a Psychiatric Treatment Order
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Required number of subjects to be included could not be accomplished
Sponsor: UMC Utrecht (Other)
Collaborators: FPC De Kijvelanden, Poortugaal (Unknown)
Responsible Party: Principal Investigator, R.L. van Ojen, MD PhD psychiatrist, UMC Utrecht
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 05/187-E
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Psychotic Disorders; Antisocial Personality Disorder; Impulse Regulation Disorder; Intermittent Explosive Disorder
MeSH Terms: conditions — Psychotic Disorders; Antisocial Personality Disorder; Disruptive, Impulse Control, and Conduct Disorders | interventions — naratriptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): four week double blind placebo treatment phase
  Interventions: Drug: placebo
- naratriptan (Active Comparator): four week double blind experimental treatment using daily naratriptan tablets
  Interventions: Drug: naratriptan

INTERVENTIONS:
Drug: naratriptan — four weeks double blind experimental treatment using oral naratriptan
  Arms: naratriptan
Drug: placebo — four weeks double blind placebo treatment
  Arms: placebo

SUMMARY:
In a double blind randomized clinical trial with cross-over design, treatment using naratriptan will be compared to placebo within a group of 30 convicts with psychiatric disorders such as psychosis or psychopathy with repeated aggressive outbursts resistant to conventional psychopharmacologic and other psychotherapeutic treatment. Hypothesis is that addition of naratriptan to the individual treatment regime reduces aggression -and improves general outcome- as compared to addition of placebo and is well tolerated in this group and under these conditions.

DETAILED DESCRIPTION:
EFFICACY OF A TRIPTAN IN THE TREATMENT OF HOSTILITY AND AGGRESSION AMONG CONVICTS WITH A PSYCHIATRIC TREATMENT ORDER

Adriano van der Loo*, Dr. Rob van Ojen**, Prof. dr. Frank Koerselman**, Prof. Dr. Henk Nijman*, Prof. Dr. Berend Olivier***

*Forensic Psychiatric Center De Kijvelanden, Poortugaal; **University Medical Center and Rudolf Magnus Institute of Neuroscience Utrecht; ***Department of Pharmacy, Utrecht University

Background

In a large number of studies, hostility, impulsivity and aggression have been demonstrated to be associated with decreased activity of the serotonergic system (Nelson and Chiavegatto 2001). In rodents a specific role for the serotonin-1b receptor has been reported (Olivier et al. 1995) and it has been shown that specific central serotonin-1b/d agonists such as lipophilic triptans have a specific anti-aggressive effect. To date, no studies have been conducted on treatment of hostility, impulsivity or aggression among humans using a triptan.

Goal of the Study

Aim is to establish the efficacy of naratriptan, registered for the treatment of migraine, as an anti-aggressive agent in patients with refractory disorders of impulse control due to psychosis or psychopathy.

Primary question is whether or not violent behavior and aggressive incidents decrease when naratriptan is administered daily in addition to treatment as usual.

Secondary questions are:

* Does overall prognosis of the underlying condition improve with the intervention?
* Can responders be differentiated from non-responders in terms of covariants including endocrine factors and polymorphisms in areas in the genome that are involved in serotonergic neurotransmission?
* Is the triptan well tolerated in this group and in this dose-range?

Study Design

Population

The sample consists of male adult volunteers with a psychiatric disorder who have been convicted and sentenced to undergo psychiatric treatment in Forensic Psychiatric Hospital "De Kijvelanden" after having committed a violent crime and have in the previous year been involved in violent incidents at least three times in spite of comprehensive psychiatric treatment of the underlying disorder.

Intervention /Drug /Dosage

In the course of a four-week period either a naratriptan 2.5 mg. tablet or a placebo tablet will be added twice to the daily medication in a double blind randomized fashion. Subsequently, after a two-week washout, patients will cross-over towards the alternative treatment condition for another four-week period.

Endpoints

Outcome will be measured using the AVL (aggression questionnaire) and the SDAS (social dysfunction and aggression scale) after 2, 4, 6, 8, and 10 weeks of treatment. Change on the CGI (Clinical Global Impression) will be compared to baseline. As usual at the study-site, the SOAS-R (Staff Observation Aggression Scale) will be filled in in case of violent incidents and type, number and duration of restraining interventions will be registered. Also recorded will be symptoms occurring during treatment and number and cause of dropout.

Description and Estimate of Risk and Burden for Participants

Safety and tolerability of both naratriptan and placebo are very well documented. Incidence and nature of side-effects and interactions has been described to be low and relatively mild, also with frequent (daily) use of naratriptan. Patients at risk for side-effects will be excluded from the study. Drugs will be added to the usual medication of the participants. A questionnaire will be administered and blood will be collected upon inclusion in the study. Data including genotype will be processed anonymously.

ELIGIBILITY:
Inclusion Criteria:

* Patient under psychiatric treatment order for violent crime
* More than two violent incidents in the year preceding inclusion, of which at least one within the last three months
* Patient is undergoing psychiatric treatment
* Informed consent

Exclusion Criteria:

* Unable for informed consent
* Intolerance for any prescription compound
* Severe liver failure (Child-Pugh grade c) of renal failure (creatinine clearance < 15 ml/min.)
* Increased risk of coronary vasospasm: symptoms of vascular disorder (including angina pectoris), history of vascular incidents, severe HBP, ECG-abnormalities in history or at screening prior to inclusion, vascular of cardial souffles.
* History of vascular incidents, hyperlipidaemia, severe HBP, DM
* Use of vasoconstrictive agents such as ergotamine derivates including methysergide, or other triptans.
* Increased risk of serotonergic syndrome: use of irreversible MAO-blocker
* Age < 18 yr. or > 65 yr.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
number of aggressive incidents | 10 weeks
aggression scores | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Frank Koerselman, MD, PhD, Study Chair — UMC Utrecht; Rob L. van Ojen, MD, PhD, Study Director — UMC Utrecht; Henk Nijman, PhD, Study Director — FPC De Kijvelanden, Poortugaal; Berend Olivier, PhD, Study Director — Utrecht University, Dep. of Pharmacy; Adriano van der Loo, MD, Principal Investigator — FPC De Kijvelanden
Locations (1):
- FPC De Kijvelanden, Poortugaal, Netherlands